CLINICAL TRIAL: NCT01315925
Title: SEIFEM 2010: Epidemiological Survey on Possible Pre-Hospital Risk Factors for Developing Invasive Fungal Infections in Patients Affected by Acute Myeloid Leukemia
Brief Title: Pre-hospital Risk Factors for Invasive Fungal Infection
Acronym: SEIFEM 2010
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Livio Pagano, MD, Catholic University of the Sacred Heart
Other Study IDs: 751/2009
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Acute Myeloid Leukemia; Aspergillosis; Candidiasis; Mycoses
Keywords: Acute myeloid leukemia; invasive fungal infection; Aspergillosis; candidiasis
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Aspergillosis; Candidiasis; Mycoses; Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Newly disgnosed AML: Adult and pediatric patients with newly diagnosed acute myeloid leukemia, both eligible and not eligible for intensive chemotherapy. Since this is a non-interventional study, therapeutic strategies remains related to local guidelines. Will be treated as cases all patients with acute leukemia in first induction developing an Invasive Fungal Infection according to international EORTC criteria for possible/probable/proven infections. Patients who do not develop the infection will be used as a control group.

SUMMARY:
SEIFEM 2010 study is a prospective, multicenter registry designed to identify and analyze risk factors for developing an invasive fungal infection in patients with newly diagnosed Acute Myeloid Leukemia, with particular interest on pre-hospital risk factors (i.e. those related to normal activities of daily life, such as occupation, location and type of residence, consume of tobacco, alcohol and others).

DETAILED DESCRIPTION:
SEIFEM 2010:

EPIDEMIOLOGICAL SURVEY ON POSSIBLE PRE-HOSPITAL RISK FACTORS FOR DEVELOPING INVASIVE FUNGAL INFECTIONS IN PATIENTS AFFECTED BY ACUTE MYELOID LEUKEMIA

Background:

In two different multicenter surveys conducted in Italy from 1988-1997 and 1999-2003, (Invasive Fungal Infections) IFIs were found to be a frequent cause of morbidity and mortality in patients treated with conventional chemotherapies, particularly in those suffering from acute myeloid leukemia (AML).

In general, the major factors that have been recognized as influencing the likelihood of invasive fungal infection are the patient's immune status, the degree of any organ damage (e.g., mucositis), and overall microbial exposure (i.e., colonization, environment, and prior infection). Since the 1990s, different risk-stratification strategies have been evaluated in order to identify those patients who may benefit from intensive prophylactic and diagnostic measures. However, despite having similar risk profiles, only a subset of AML patients will develop an IFI. One of the most exciting recent advances in the understanding of the epidemiology of IFIs is the recognition of the complexity of the host and the identification of new host-related risk factors.

Aim of this study is to identify and analyze risk factors for developing an invasive fungal infection in patients with newly diagnosed Acute Myeloid Leukemia, with particular interest on pre-hospital risk factors.

Aims and objective:

* To identify high risk subjects that can take advantage of an antifungal prophylaxis or an early antifungal treatment (preemptive treatment).
* To identify possible fungal infections sources for the period preceding the diagnosis of leukemia, in particular those related to normal activities of daily life (e.g. occupation, location and type of residence, consume of tobacco, alcohol or illicit drugs and others).
* To analyze hospital-related sources of fungal infection, from well known predisposing factors (i.e. duration and severity of neutropenia) to other like central venous catheter, urinary catheter, comorbidities, etc.
* To analyze the impact of both the prophylactic regimen adopted and the antifungal treatment.

Design:

* Prospective, multicenter, observational and clinical-epidemiological study.
* The study is expected to enroll at least 500 patients with newly diagnosed acute myeloid leukemia, those eligible for treatment and those not eligible, within 2 years or until the achievement of a statistically evaluable number of cases.
* SEIFEM 2010 is a noninterventional registry and therefore there will not be any any change physicians' diagnostic and therapeutic choices, that remain related to local guidelines.
* Every patient who accept to take part to the study, will be asked to read and sign an informed consent.
* An apposite form, with a detailed epidemiological section, should be compiled by clinicians for each enrolled patient.
* A complete information page on the study is supplied to each patient enrolled.

Data collection:

In the questionnaire, possible risk factors for invasive fungal infections, prior to the onset of acute leukemia, are evaluated. The module consists of several sections:

* Personal information (age, sex, observation time of the case, AML subtype, performance status at admission), patient data will be anonymous.
* Comorbidities (diabetes, chronic renal failure, COPD, chronic liver disease, previous TBC)
* A section compiled by the patient about possible risk factors related to the daily living habits (location and type of residence, profession, hobbies, pets, personal hygiene, ambiental exposures, consume of tobacco, alcohol or illicit drugs and others)
* A second part of the form will be compiled at the time of evaluation after induction chemotherapy (between 30 and 40 days after chemotherapy) or, for those not suitable for conventional treatment, 30-40 days after diagnosis.

At the time of a diagnosis of fungal infection data on the type of infection, treatment and course of infection will be evaluated.

Eligibility:

Adult and pediatric patients with newly diagnosed acute myeloid leukemia, both eligible and not eligible for intensive chemotherapy. Since this is a noninterventional study, therapeutic strategies remains related to local guidelines. Will be treated as cases all patients with acute leukemia in first induction developing an Invasive Fungal Infection according to international EORTC criteria for possible/probable/proven infections. Patients who do not develop the infection will be used as a control group.

Participating centers:

Forty-three Italian divisions of Hematology will take part to the study, distributed among universities and highly specialized hospitals located throughout the country.

ELIGIBILITY:
Inclusion Criteria:

* all newly diagnosed AML who accept to take part to the registry and sign an informed consent

Exclusion Criteria:

* relapsing/refractory AML
* patients who do not sign informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric patients with newly diagnosed acute myeloid leukemia, both eligible and not eligible for intensive chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-01

PRIMARY OUTCOMES:
Incidence of Invasive fungal infections | 30th day after the end of first line chemotherapy
  To identify possible fungal infections sources for the period preceding the diagnosis of leukemia, in particular those related to normal activities of daily life (e.g. occupation, location and type of residence, consume of tobacco, alcohol or illicit drugs and others).

CONTACTS AND LOCATIONS:
Locations (42):
- Italy (42):
  - University of Ancona, Ancona, AN
  - University of Bary, Bari, BA
  - University of Bologna, Bologna, BO
  - Catholic University, Campobasso, Campobasso
  - University of Firenze, Florence, FI
  - Tricase Hospital, Tricase, LE
  - Niguarda Hospital, Milan, MI
  - Catholic University, Rome, RM
  - IFO, Rome, RM
  - S.Camillo Hospital, Rome, RM
  - S.Giovanni Hospital, Rome, RM
  - University of Tor Vergata, Rome, RM
  - Le Molinette Hospital, Torino, TO
  - Hospital of Brescia, Brescia
  - University of Cagliari, Cagliari
  - Cuneo Hospital, Cuneo
  - Istotuto Meyer, Florence
  - Gaslini Hospital, Genova
  - La Spezia Hospital, La Spezia
  - Lecce Hospital, Lecce
  - Lecce Pediatric Hospital, Lecce
  - University of Modena e Reggio, Modena
  - Monza Hospital, Monza
  - San Gerardo Hospital, Monza
  - "Federico II" University, Napoli
  - Cardarelli Hospital, Napoli
  - Pausilion Hospital, Napoli
  - University of Palermo, Palermo
  - University of Parma, Parma
  - S.Matteo Hospital, Department of Hematology, Pavia
  - S.Matteo Hospital, Department of Medicine, Pavia
  - University of Perugia, Pediatric Hematology, Perugia
  - University of Perugia, Perugia
  - Pescara Hospital, Pescara
  - Reggio Calabria Hospital, Reggio Calabria
  - Reggio Emilia Hospital, Reggio Emilia
  - "Padre Pio" Hospital, San Giovanni Rotondo
  - Regina Margherita Hospital, Torino
  - S.Anna Hospital, Torino
  - University of Udine, Udine
  - University of Verona, Verona
  - Verona Hospital, Verona

REFERENCES:
- [Background] Caira M, Mancinelli M, Leone G, Pagano L. Invasive aspergillosis in acute leukemias: old and new risk factors and epidemiological trends. Med Mycol. 2011 Apr;49 Suppl 1:S13-6. doi: 10.3109/13693786.2010.509138. Epub 2010 Aug 26. PMID 20795761
- [Background] Muhlemann K, Wenger C, Zenhausern R, Tauber MG. Risk factors for invasive aspergillosis in neutropenic patients with hematologic malignancies. Leukemia. 2005 Apr;19(4):545-50. doi: 10.1038/sj.leu.2403674. PMID 15729382
- [Background] Pagano L, Caira M, Candoni A, Offidani M, Martino B, Specchia G, Pastore D, Stanzani M, Cattaneo C, Fanci R, Caramatti C, Rossini F, Luppi M, Potenza L, Ferrara F, Mitra ME, Fadda RM, Invernizzi R, Aloisi T, Picardi M, Bonini A, Vacca A, Chierichini A, Melillo L, de Waure C, Fianchi L, Riva M, Leone G, Aversa F, Nosari A. Invasive aspergillosis in patients with acute myeloid leukemia: a SEIFEM-2008 registry study. Haematologica. 2010 Apr;95(4):644-50. doi: 10.3324/haematol.2009.012054. Epub 2009 Oct 22. PMID 19850903
- [Derived] Caira M, Candoni A, Verga L, Busca A, Delia M, Nosari A, Caramatti C, Castagnola C, Cattaneo C, Fanci R, Chierichini A, Melillo L, Mitra ME, Picardi M, Potenza L, Salutari P, Vianelli N, Facchini L, Cesarini M, De Paolis MR, Di Blasi R, Farina F, Venditti A, Ferrari A, Garzia M, Gasbarrino C, Invernizzi R, Lessi F, Manna A, Martino B, Nadali G, Offidani M, Paris L, Pavone V, Rossi G, Spadea A, Specchia G, Trecarichi EM, Vacca A, Cesaro S, Perriello V, Aversa F, Tumbarello M, Pagano L; SEIFEM Group (Sorveglianza Epidemiologica Infezioni Fungine in Emopatie Maligne). Pre-chemotherapy risk factors for invasive fungal diseases: prospective analysis of 1,192 patients with newly diagnosed acute myeloid leukemia (SEIFEM 2010-a multicenter study). Haematologica. 2015 Feb;100(2):284-92. doi: 10.3324/haematol.2014.113399. PMID 25638805
- [Derived] Pagano L, Verga L, Busca A, Martino B, Mitra ME, Fanci R, Ballanti S, Picardi M, Castagnola C, Cattaneo C, Nadali G, Nosari A, Candoni A, Caira M, Salutari P, Lessi F, Aversa F, Tumbarello M. Systemic antifungal treatment after posaconazole prophylaxis: results from the SEIFEM 2010-C survey. J Antimicrob Chemother. 2014 Nov;69(11):3142-7. doi: 10.1093/jac/dku227. Epub 2014 Jun 19. PMID 24948702
- [Derived] Pagano L, Caira M, Candoni A, Aversa F, Castagnola C, Caramatti C, Cattaneo C, Delia M, De Paolis MR, Di Blasi R, Di Caprio L, Fanci R, Garzia M, Martino B, Melillo L, Mitra ME, Nadali G, Nosari A, Picardi M, Potenza L, Salutari P, Trecarichi EM, Tumbarello M, Verga L, Vianelli N, Busca A; SEIFEM Group. Evaluation of the practice of antifungal prophylaxis use in patients with newly diagnosed acute myeloid leukemia: results from the SEIFEM 2010-B registry. Clin Infect Dis. 2012 Dec;55(11):1515-21. doi: 10.1093/cid/cis773. Epub 2012 Sep 5. PMID 22955439